CLINICAL TRIAL: NCT03167944
Title: "Comparison of Traditional Electrosurgery System Versus Low Thermal Tissue Dissection System for Total Mastectomy: A Prospective Randomized Controlled Trial"
Brief Title: Traditional Electrosurgery System Versus Low Thermal Tissue Dissection System for Total Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suebwong Chuthapisth, Asst. Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: convplas
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Seroma
Keywords: Mastectomy; Seroma
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional electrocautery (Experimental)
  Interventions: Device: Conventional Electrocautery
- Low thermal electrosurgery system (Experimental)
  Interventions: Device: Low thermal electrosurgery system

INTERVENTIONS:
Device: Low thermal electrosurgery system — PEAK Plasmablade
  Arms: Low thermal electrosurgery system
Device: Conventional Electrocautery — Conventional Electrocautery
  Arms: Conventional electrocautery

SUMMARY:
Breast cancer is one of the most common cancer among women nowadays. There are lots of modality of treatment and one of them is Mastectomy. We found out that seroma is one of the disturbing postoperative complications after mastectomy. In our study we want to compare the outcome between using the conventional electrocautery and the low thermal tissue dissection. We expected that the serum production should be lower in cases using low thermal system electrosurgery system.

ELIGIBILITY:
Inclusion Criteria:

* Female aged >18 years old
* Patients that fulfill the indication of mastectomy
* Medium-sized breast volume (Breast weight < 1500 grams)

Exclusion Criteria:

* Patients who cannot complete the informed consent
* Patients with ASA CLASS > 3

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-03-25 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Drainage volume after surgery | Up to 24 weeks
  Drainage volume detected after surgery which is measured in drainage container and measured by syringe gauge aspiration

SECONDARY OUTCOMES:
Post operative Pain | Up to 24 weeks
  Post-operative Pain measured using 0-10 Numeric pain scale
Patient's Hospital costs | up to 1 week
  Expenses that the patient has to pay while staying in the hospital
Wound infection | Up to 24 weeks
  Wound infection after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Bangkok, Thailand